CLINICAL TRIAL: NCT02884934
Title: Six Years of Follow-up After Extended Duration of Oral Anticoagulant Therapy for a First Episode of Idiopathic Pulmonary Embolism or Proximal Deep Vein Thrombosis.
Brief Title: Six Years of Follow-up After Idiopathic Venous Throbmoembolism
Acronym: Padis-Ext
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: Padis-Extension (RB 12.075)
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Last update posted 2025-03-21 (Actual); Status verified 2025-02

CONDITIONS: Pulmonary Embolism; Proximal Deep Vein Thrombosis
Keywords: venous thromboembolism; recurrent venous thromboembolism; anticoagulant-related bleeding
MeSH Terms: conditions — Pulmonary Embolism; Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Beyond the first 6 months of anticoagulation, patients with a first episode of unprovoked venous thromboembolism have a high risk of recurrence after stopping anticoagulations. Extending anticoagulant therapy for an additional 18 months is associated with a major reduction of recurrent VTE; however this benefit tended to be lost after stopping anticoagulation during a follow-up period of two years. This risk of recurrentce is likely to continuously increase over the years as well as the risk of chronic thromboembolic pulmonary hypertension (after pulmonary embolism) or the risk of post-thrombotic syndrome (after deep vein thrombosis). The aim of the PADIS-EXTENSION trial is to estimate these risks over 6 years of follow-up in patients who have been initially treated during 6 months or 24 months (patients included in the PADIS PE and PADIS DVT trial).

DETAILED DESCRIPTION:
Beyond the first 6 months of anticoagulation, patients with a first episode of unprovoked venous thromboembolism have a high risk of recurrence after stopping anticoagulations (about 10% at one year and 30% at 5 years). Extending anticoagulant therapy for an additional 18 months is associated with a major reduction of recurrent VTE; however this benefit tended to be lost after stopping anticoagulation during a follow-up period of two years. This has been well demonstrated in the double-blind randomized PADIS PE trial comparing 2 years with 6 months of anticoagulation and a follow-up of two years after study treatment discontinuation. This risk of recurrence is likely to continuously increase over the years as well as the risk of chronic thromboembolic pulmonary hypertension (after pulmonary embolism) or the risk of post-thrombotic syndrome (after deep vein thrombosis). In addition, risk factors of such complications remain uncertain. The first aim of the PADIS-EXTENSION trial is to estimate these risks over 6 years of follow-up in patients who have been initially treated during 6 months or 24 months (patients included in the PADIS PE and PADIS DVT trial). Secondary aims are to identify risk factors of these complications during long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a first episode of idiopathic pulmonary embolism or idiopathic proximal deep vein thrombosis who have been initially treated during 6 months or 24 months using Vitamin K antagonist with a INR between 2 and 3 and enrolled in clinical study Padis-Ep and Padis TVP

Exclusion Criteria:

Participation refused

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: idiopathic pulmonary embolism /Idiopathic Proximal Deep Vein Thrombosis
Sampling Method: Probability Sample
Enrollment: 409 (Actual)
Dates: Start 2013-03-28 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
Symptomatic recurrent venous thromboembolism | 6 years

SECONDARY OUTCOMES:
Major Bleeding | 6 years
Chronic Thromboembolic Pulmonary Hypertension | 6 years
Post-Thrombotic Syndrome | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Francis COUTURAUD, Study Director — CHRU de Brest
Locations (10):
- France (10):
  - CHRU de Brest, Brest
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Grenoble, Grenoble
  - CH de Lannion, Lannion
  - CH de Lorient, Lorient
  - Hôpital Européen Georges Pompidou, Paris
  - CHU de Rennes, Rennes
  - CH St Brieuc, Saint-Brieuc
  - CHU de St Etienne, Saint-Etienne
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided